CLINICAL TRIAL: NCT00061529
Title: A Phase III Study of Brimonidine Tartrate Ophthalmic Solution, 0.15% in Patients With Open-Angle Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-02-49
Record Dates: First submitted 2003-05-28; First posted 2003-05-30 (Estimated); Last update posted 2008-08-05 (Estimated); Status verified 2008-08

CONDITIONS: Open-Angle Glaucoma; Ocular Hypertension
Keywords: Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

INTERVENTIONS:
Drug: Brimonidine Tartrate Ophthalmic Solution

SUMMARY:
The primary objective of this study is to compare the safety and efficacy of Brimonidine Tartrate Ophthalmic Solution, 0.15% in patients with open-angle glaucoma or ocular hypertension.

ELIGIBILITY:
* Patients of any race
* two (2) years of age or older
* of either sex
* diagnosed with open-angle glaucoma (with or without pseudoexfoliation or pigment dispersion component)or ocular hypertension

Min Age: 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-01; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Alcon Call Center, Fort Worth, Texas, United States